CLINICAL TRIAL: NCT03983759
Title: Clinical Study of Sequential Sequential Sintilimab Maintenance Therapy in Patients With Extensive Small Cell Lung Cancer After Chemotherapy Combined With Adoptive Cellular Immunotherapy
Brief Title: Study of Sintlimab Maintenance Therapy in Patients With Extensive Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH immunotherapy002
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2019-06

CONDITIONS: Small Cell Lung Cancer; Extensive Disease; Adoptive Cellular Immunotherapy; Chemotherapy; Maintenance
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): phlebotomation 50ml 1-7 days before chemotherapy for culture of R-CIK cells chemotherapeutic regimen EP or EC as follows: VP-16 100mg/m2 D1-3 plus cisplatin 75mg/m2 D1 or VP-16 100mg/m2 D1-3 plus carboplatin AUC=5 D1 R-CIK cells were transfused back to the patients 2-7 days after the end of chemotherapy, and the amount of R-CIK cells returned each time was about 5×109 three weeks each cycle efficacy evaluated every two cycles patients with the efficay is CR, PR or SD after 4-6 cycles enter the sintilimab maintenance therapy for one year or until the progression of disease, or occurrence of intolerable adverse events.
  the dose of sintilimab is fixed dose of 200mg every three weeks
  Interventions: Drug: sintilimab maintenance

INTERVENTIONS:
Drug: sintilimab maintenance — the patients with CR, PR or SD after the chemotherapy plus R-CIK will receive sintilimab maintenance therapy. The dose of sintilimab is fixed at 200mg every three weeks.

SUMMARY:
Small cell lung cancer is a highly aggressive malignancy. Currently, there is no effective regimen for patients after the progression offirst-line chemotherapy. The prognosis of patients with extensive disease is very poor, and the improved therapeutic efficacy is urgently needed. Most patients with small cell lung cancer have a long history of smoking, and the tumor mutation burden is relatively high, which provides potential for immunological checkpoint inhibitors represented by PD-1 antibodies. A number of studies have shown that chemotherapy combined with adoptive cellular immunotherapy could prolong the survival of patients. This study is a clinical study to explore the efficacy and safety of maintenance therapy with sintilimab after 4-6 cycles of first-line chemotherapy combined with adoptive cellular immunotherapy in patients with advanced small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* small cell lung cancer confirmed by pathology
* extensive small cell lung cancer by imaging
* at least one measurable lesion by RECIST 1.1
* ECOG 0-1
* adequate organ function
* no other severe diseases conflicting with this regimen (such as autoimmune diseases, immunodeficiency, organ transplantation, etc)
* no history of other maliganancies
* Women of childbearing period must examinate for a negative pregnancy test within 7 days, use appropriate contraceptive measures during the study and 6 months after the trial.
* agreement to participate in the study and signed informed consent from the patients

Exclusion Criteria:

* serious infectious diseases four weeks before enrollment
* requirement intermittent use of bronchodilators or medical interventions;
* the use of immunosuppressants before the enrollment, the amount of immunosuppressant used ≥10mg / day oral prednisone for more than 2 weeks;
* severe allergies
* severe mental disorders
* abnormal coagulation function
* previous or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, severe lung damage, etc.
* other situations considered by investigators not meet the inclusion criteria (including but not limited to symptomatic brain metastases)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
median survival time | two years.
  the period from the day of enrollment to the date of death

SECONDARY OUTCOMES:
progression-free survival | six months
  the period from the day of enrollment to the date of confirmed progression or death depending on which one occurs first.
objective response rate of sintilimab | six month
  from the date of first dose of sintilimab to the date of confirmed progression following
adverse events rate of sintilimab | one year
  the rate of adverse events during the maintenance therapy of sintilimab

CONTACTS AND LOCATIONS:
Overall Officials: Jing Ding, Master, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma B, Zhou Y, Shang Y, Zhang Y, Xu B, Fu X, Guo J, Yang Y, Zhang F, Zhou M, Huang H, Li F, Lin H, Zhao L, Wang Z, Gao Q. Sintilimab maintenance therapy post first-line cytokine-induced killer cells plus chemotherapy for extensive-stage small cell lung cancer. Front Oncol. 2022 Sep 9;12:852885. doi: 10.3389/fonc.2022.852885. eCollection 2022. PMID 36158690